CLINICAL TRIAL: NCT02987283
Title: Safer Sleep: A Diagnostic Accuracy Study Evaluating Breath Sound Recordings and STOP-Bang In Screening For Obstructive Sleep Apnea While Awake
Brief Title: Evaluating Accuracy of Breath Sound Recordings and STOP-Bang Screening For Obstructive Sleep Apnea While Awake
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Other Study IDs: REB 2016-0494
Record Dates: First submitted 2016-05-25; First posted 2016-12-08 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will perform a diagnostic accuracy study comparing tracheal breath sound recordings in awake individuals to the STOP-Bang screening questionnaire, using the apnea-hypopnea index (AHI) score determined by polysomnography as the gold standard.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a breathing disorder with numerous health effects including a greater risk of peri-operative anesthetic complications. Numerous screening tools exist but are not without limitations. Diagnostic overnight sleep studies are resource-intensive and difficult to obtain in the short time period between pre-operative clinic assessment and the day of surgery.

This project aims to test the diagnostic performance of a new screening technology, Awake-OSA, for screening of obstructive sleep apnea (OSA). "Awake-OSA" uses a small external microphone placed on the neck, to record and analyze tracheal breath sounds at the bedside while the patient is awake.

Using polysomnography (PSG) as a gold standard, the investigators will compare Awake-OSA (breath sound recording) and the STOP-Bang screening questionnaire in their ability to accurately identify patients with OSA, as well as classify OSA in terms of severity.

Early, point-of-care diagnosis has the potential to provide a low-cost, convenient alternative to traditional screening questionnaires and enable more selective use of PSG. Our goal is to improve peri-operative patient safety while improving use of resources and streamlining patient care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older.
* Referred for diagnostic sleep study.
* Willing and able to consent.

Exclusion Criteria:

* Under the age of 18 yrs.
* Unwilling or unable to give consent.
* Expected to have an abnormal EEG (epilepsy, brain tumour, deep brain stimulator).
* Significant craniofacial abnormality (ex. unrepaired cleft lip/palate).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort will be selected from patients referred to the Ottawa Hospital sleep clinic for a diagnostic sleep study.
Sampling Method: Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-09-20 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Screening and diagnostic test performance of Awake-OSA and STOP-Bang | Night 1
  Screening and diagnostic test performance of Awake-OSA and STOPBang in identifying OSA vs non-OSA patients, using AHI as gold-standard reference.

SECONDARY OUTCOMES:
Development of new diagnostic algorithm determined by predictive values, sensibility, and specificity | Through study completion, average two years
  The investigators will calculate positive and negative predictive values, sensibility, and specificity or each diagnostic tool tested in the study as well as for a combination of these tools to determine the best possible diagnostic algorithm for OSA. Positive and negative predictive values, sensibility, and specificity of the resulting diagnostic algorithm will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Boet, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided